CLINICAL TRIAL: NCT06983808
Title: The PREBEAT Trial: Digital PREhaBilitation in thE Cardiac Surgical populATion
Acronym: PREBEAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claire Hines (Other)
Collaborators: Melbourne Health (Other)
Responsible Party: Sponsor-Investigator, Claire Hines, Site Investigator, RMIT University
Organization: RMIT University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RMIT-HREC 28861; RMH-HREC 2024.163 (Other: Royal Melbourne Hospital)
Record Dates: First submitted 2025-04-30; First posted 2025-05-21 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Digital Health; Telehealth; CABG; Cardiac Surgery; Heart Surgery; Prehabilitation; Perioperative
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Masking Description: Surgeons and Hospital Ward Staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients in this arm receive standard preparation for surgery as per hospital procedure. This may include information sessions, pamphlets, and meetings with clinicians.
  Interventions: Other: Control (Standard treatment)
- Digital Health Arm (Experimental): Patients in this arm engage in digital health prehabilitation which involves exercise, nutrition and information and scheduled telehealth to assist with preparation for surgery.
  Interventions: Other: Digital Cardiac Prehabilitation

INTERVENTIONS:
Other: Digital Cardiac Prehabilitation — Digital Cardiac Prehabilitation - A combined telehealth and app-based preparation for cardiac surgery
  Arms: Digital Health Arm
Other: Control (Standard treatment) — Standard preparation for surgery as per Melbourne Health hospital procedures and processes. This may include information sessions, pamphlets, and meetings with clinicians. This does not include a prehabilitation program.
  Arms: Control

SUMMARY:
The goal of this randomised controlled trial is to learn if a digital prehabilitation program is feasible in patients awaiting cardiac surgery. The main questions it aims to answer are:

1. Is the digital health program usable?
2. Is the digital health program acceptable?
3. Do patients adhere to the digital health program?

Researchers will compare a group using the digital prehabilitation program with standard care to see if the program is feasible and explore any differences in health outcomes.

Participants will

* Use a digital health mobile phone application to guide you through exercise, nutrition and preparation for surgery.
* Engage in telehealth consultations.
* Complete questionnaires
* Complete exercise testing

ELIGIBILITY:
Inclusion Criteria:

* 21 days+ prior to cardiac surgery
* Able to provide consent,
* Proficient in English to understand questionnaires, training instructions and outcome assessments.
* Digitally literate to independently navigate a smart device and novel application.

Exclusion Criteria:

* severe or unstable neurological, cardiorespiratory, or musculoskeletal disease or mental illness that might compromise ability to perform exercise,
* unstable psychiatric or cognitive disorders,

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Usability of Digital Cardiac Prehabilitation as assessed by the Mhealth Application Usability Questionnaire (MAUQ) | 2 days Pre-operatively
  mAUQ is an 18-item questionnaire for patients to evaluate the usability of the digital application under the three domains of; Ease of Use, Interface, Satisfaction and Usefulness.
  Low numbers indicate a higher perception of usability with the digital interface for participants.
Adherence of Digital Cardiac Prehabilitation as measured by usage metrics from Mobile Phone App metrics | 2 days Pre-operatively
  Metrics Used include
  * Time and date: when the application is accessed.
  * Dwell Time: how much time is spent on a particular page.
  * Number of pages viewed: how many views per page per day.
  * User input data: data the user submits in the app, including minutes walked, exercises marked as complete, and questionnaires completed.
Acceptability of Digital Cardiac Prehabilitation as measured by Theoretical Framework of Acceptability Questionnaire (TFA) | 2 days Pre-operatively
  TFA-Q is composed of eight items, in alignment with the eight acceptability constructs (Affective attitude, Burden, Ethicality, Perceived effectiveness, intervention coherence, self-efficacy, opportunity costs, general acceptability).
  High numbers indicate a more acceptable digital experience.
Incidence of Adverse events | Recorded through study completion, an average of 7 months.
  Adverse events, defined as any undesirable event, such as injury, fall, and discomfort related to prehabilitation will be recorded and severity will be reported according to hospital policy.
  Lower numbers are more favourable, indicating fewer adverse events.

SECONDARY OUTCOMES:
Health service use as measured by Length of Stay (LOS) | 30 days post-operatively
  Hospital services use measured by length of stay (LOS) (days) - gained using hospital administrative data.
  Low numbers are preferable, indicating the patient has not stayed as long in hospital.
Health service use as measured by Intensive Care Unit (ICU) Length of Stay (ICU LOS) | 30 days post-operatively
  Hospital services use as measured by ICU LOS (days), gained using hospital administrative data.
  Low numbers are preferable, indicating the patient has not required as intensive care.
Health service use as measured by Readmissions | 30 days post-operatively
  Hospital services use as measured by the incidence of Readmissions, gained using hospital administrative data.
  Low numbers are preferable, indicating the patient has had less need to return to hospital for care, following discharge.
Health service use as measured by the Health Utilization Questionnaire (HUQ) | Post operatively at Time Points: 2 weeks, 30 days, 3 months and 6 months
  The HUQ is 12 item survey which assesses the frequency and type of healthcare services accessed by individuals. It gathers data on medical visits, hospital stays, medication use, and other healthcare interactions to evaluate healthcare consumption, and includes modern communication systems of engaging with health care services.
  Low numbers are preferable, indicating less need to engage with health services.
Mortality as measured by days alive out of hospital (DAoH) | 6 months post-operatively
  Mortality as measured by days alive out of hospital. This data will be gained using hospital administrative records in the event that the patient is uncontactable.
  DAoH should be equal to the number of days since discharge. Where DAoH are lower than the number of days since discharge, this is less favourable, indicating the patient has not survived.
Cost of program delivery as estimated by multiplying the occasions of service by relevant national average hospital award wages for respective staff. | 6 months post-operatively
  Hospital administrative records will be used to supplement resource use data from surveys on consent from participants. In addition, the lead patient-facing researcher will maintain a clinician log, documenting time spent with each patient during the intervention phase to accurately represent the equivalent cost of the intervention. This is expected to include time used for adjusting or maintaining physical activity programs, and any interactions online, via phone, or telehealth. Cost of program delivery will be calculated on conclusion of the PREBEAT trial.
  Low cost is preferable, indicating a potential financial benefit to health services which provide prehabilitation programs.
Recovery as measured by the Post-Operative Quality of Recovery Scale (PostopQRS). | Baseline, 2 days pre-operatively, Post operatively at Time Points: 1 day, 3 days, day of discharge, 2 weeks, 30 days, 3 months and 6 months.
  Recovery will be assessed using the 5-domain the Post-Operative Quality of Recovery Scale (PostopQRS). This scale has been designed to quantify quality of recovery ((physiological, emotive, nociceptive, activities of daily living, cognitive and patient perspective) after surgery and anaesthesia. It is comprised of questions that objectively measure patient recovery over multiple time periods. This assessment has been validated and used extensively in the cardiac surgical population. The PostopQRS will be used to monitor multidomain recovery at pre and post intervention timepoints, postoperatively and throughout recovery.
Functional outcome as measured by the Functional Difficulties Questionnaire shortened (FDQs) | Baseline, 2 days pre-operatively, Post operatively at day of discharge, 2 weeks, 30 days, 3 months and 6 months.
  The Functional Difficulties Questionnaire shortened (FDQs) is a 10-item functional outcome measure which asks the participant to rate the difficulty they experience when completing a series of 10 upper limb and trunk activities by placing a mark along a 10cm line, with anchors indicating "no difficulty" and "maximum difficulty". For those activities that participants could not attempt whilst completing the questionnaire due to the institution sternal precautions, they are asked to think back to the last time they performed the task.
  Individual scores, measured to the nearest centimetre (cm), are aggregated to form a total out of 130 with higher scores representing greater difficulty experienced during functional activities.
Body metrics as measured by Body Mass Index (BMI) | Baseline, 3 months post-operatively.
  Height (cm) and weight (kg) are taken and placed into the formula: BMI = weight (kg) / [height (m)]². BMI healthy range is 18.5-24.9, with patients being above this overweight (or obese if over 30).
Body metrics as measured by Waist Hip Ratio (WHR) | Baseline, 3 months post-operatively.
  Waist and hip measurements (cm) are taken and placed into the formula: WHR= waist circumference / hip circumference. Higher numbers of WHR (above 0.85 in women, and 0.99 in men) indicate a higher risk factor for development of some chronic diseases.
Body composition (Bioimpedance) as measured by non-invasive tetrapolar bioimpedance spectroscopy (BIS, SOZO, Impedimed, USA). | Baseline, 3 months post-operatively.
  Bioimpedance will be measured by non-invasive tetrapolar bioimpedance spectroscopy (BIS, SOZO, Impedimed, USA), used for estimating body composition (including muscle mass) by determining the resistance to the flow of an electrical current through body water.
  Increases in lean muscle percentages can indicate positive adaptations to exercise.
Postoperative pulmonary complications (PPCs) as measured the Melbourne Group Score (MGS) | Post operatively at Time Points: 1 day, 3 days, day of discharge.
  The Melbourne Group Score (MGS) is a clinical tool used to diagnose postoperative pulmonary complications (PPCs) in patients following surgery. It consists of a set of criteria including abnormal chest x-ray, fever, elevated white cell count, production of purulent sputum, positive respiratory culture, oxygen saturation below 90% on room air, and clinical signs of pulmonary infection.
  If a patient has the presence of four or more criteria in a 24-hour period it is diagnostic of a PPC.
  Lower numbers of PPC through the study are preferable, indicating a lower number of chest infections.
Functional capacity as measured by 1-Minute Sit-to-Stand (1STS) | Baseline, 2 days pre-operatively, Post operatively at day of discharge, 3 months and 6 months.
  The 1-Minute Sit-to-Stand (1STS) assessment is a simple, quick test used to evaluate lower body strength, endurance, and functional capacity. The participant is asked to stand up from a seated position and sit back down as many times as possible within one minute. The total number of repetitions is recorded as the score.
  Higher scores indicate a better functional capacity.
Inspiratory muscle strength as measured by Maximal Inspiratory Pressure (MIP) | Baseline, 2 days pre-operatively, and 3 months post-operatively.
  Maximal Inspiratory Pressure (MIP) is a measure of inspiratory muscle strength and will be measured via a maximal inspiratory effort using the Powerbreathe KH2. Patients will be asked to sit comfortably in a chair with their feet flat on the ground, with a nose clip on. Patient's will be asked to completely exhale, then form a secure lip seal around the mouthpiece and inhale as forcefully as possible through the device. The KH2 Powerbreathe will measure the pressure generated during this maximal inspiratory effort. This process will be repeated twice, with a 1-minute rest between efforts. The highest pressure generated will be recorded as the patient's MIP.
  Higher pressures are preferable, indicating stronger inspiratory muscles.
Adherence to the Mediterranean diet as measured by The MEDAS (Mediterranean Diet Adherence Screener) | Baseline, 2 days pre-operatively, Post operatively at day of discharge, 30 days, 3 months and 6 months.
  The MEDAS (Mediterranean Diet Adherence Screener) is a 14-item questionnaire designed to evaluate adherence to the Mediterranean diet. Each item assesses the frequency or amount of specific food consumption or dietary habits associated with the Mediterranean diet, such as olive oil, fruits, vegetables, nuts, fish, legumes, and wine. Points are assigned for each item, with higher scores indicating greater adherence to the diet.
Anxiety as measured by The State-Trait Anxiety Inventory (STAI) | Baseline, 2 days pre-operatively, Post operatively at the day of discharge, 2 weeks, 30 days, 3 months and 6 months.
  The State-Trait Anxiety Inventory (STAI) is a 40 item psychological assessment tool that measures anxiety in adults and is commonly used in prehabilitation research. It distinguishes between two types of anxiety: state anxiety (a temporary condition experienced in specific situations) and trait anxiety (a general tendency to respond with anxiety across many situations). To reduce the patient assessment burden, the shorted version: State-Trait Anxiety Inventory (STAI-6) will be used in this study.
  Lower scores are preferable, indicating a less anxious patient.
Self-Efficacy as measured by The General Self-Efficacy Scale (GSE) | Baseline, 2 days pre-operatively, Post operatively at the day of discharge, 2 weeks, 30 days, 3 months and 6 months.
  The General Self-Efficacy Scale (GSE) is a 10-item questionnaire designed to assess an individual's belief in their ability to handle various stressful situations and challenges. Each item is rated on a 4-point Likert scale, ranging from "Not at all true" to "Exactly true." Higher scores indicate greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Royse, MD - Cardiothoracic Surgeon, Principal Investigator — Melbourne Health
Locations (1):
- Melbourne Health (Royal Melbourne and Melbourne Private Hospital), Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data summary from primary and secondary outcome measures
Supporting Information: Study Protocol, ICF
Time Frame: By at least Jan 2027, for at least 12 months.
Access Criteria: By Journal Article Publication and/or conference posters, proceedings and/or presentations.

REFERENCES:
- [Background] Steinmetz C, Bjarnason-Wehrens B, Walther T, Schaffland TF, Walther C. Efficacy of Prehabilitation Before Cardiac Surgery: A Systematic Review and Meta-analysis. Am J Phys Med Rehabil. 2023 Apr 1;102(4):323-330. doi: 10.1097/PHM.0000000000002097. Epub 2022 Sep 23. PMID 36149383
- [Background] Doyle MP, Indraratna P, Tardo DT, Peeceeyen SC, Peoples GE. Safety and efficacy of aerobic exercise commenced early after cardiac surgery: A systematic review and meta-analysis. Eur J Prev Cardiol. 2019 Jan;26(1):36-45. doi: 10.1177/2047487318798924. Epub 2018 Sep 6. PMID 30188177
- [Background] Kehler DS, Stammers AN, Tangri N, Hiebert B, Fransoo R, Schultz ASH, Macdonald K, Giacomontonio N, Hassan A, Legare JF, Arora RC, Duhamel TA. Systematic review of preoperative physical activity and its impact on postcardiac surgical outcomes. BMJ Open. 2017 Aug 11;7(8):e015712. doi: 10.1136/bmjopen-2016-015712. PMID 28801404
- [Background] Magon A, Caruso R, Sironi A, Mirabella S, Dellafiore F, Arrigoni C, Bonavina L. Trajectories of Health-Related Quality of Life, Health Literacy, and Self-Efficacy in Curatively-Treated Patients with Esophageal Cancer: A Longitudinal Single-Center Study in Italy. J Patient Exp. 2021 Nov 29;8:23743735211060769. doi: 10.1177/23743735211060769. eCollection 2021. PMID 35252557
- [Background] Nijkamp MD, Kenens CA, Dijker AJ, Ruiter RA, Hiddema F, Nuijts RM. Determinants of surgery related anxiety in cataract patients. Br J Ophthalmol. 2004 Oct;88(10):1310-4. doi: 10.1136/bjo.2003.037788. PMID 15377557
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Hulzebos EH, van Meeteren NL, van den Buijs BJ, de Bie RA, Brutel de la Riviere A, Helders PJ. Feasibility of preoperative inspiratory muscle training in patients undergoing coronary artery bypass surgery with a high risk of postoperative pulmonary complications: a randomized controlled pilot study. Clin Rehabil. 2006 Nov;20(11):949-59. doi: 10.1177/0269215506070691. PMID 17065538
- [Background] Birrer DL, Kuemmerli C, Obwegeser A, Liebi M, von Felten S, Pettersson K, Horisberger K. INSPIRA: study protocol for a randomized-controlled trial about the effect of spirometry-assisted preoperative inspiratory muscle training on postoperative complications in abdominal surgery. Trials. 2022 Jun 7;23(1):473. doi: 10.1186/s13063-022-06254-4. PMID 35672861
- [Background] Beaujolin, A., Mané, J., Presse, C., Barbosa-Silva, J., Bernini, M., Corbellini, C., & De Abreu, R. M. (2024). Inspiratory Muscle Training Intensity in Patients Living with Cardiovascular Diseases: A Systematic Review. Hearts, 5(1), 75-90.
- [Background] Patsaki I, Kouvarakos A, Vasileiadis I, Koumantakis GA, Ischaki E, Grammatopoulou E, Kotanidou A, Magira EE. Low-Medium and High-Intensity Inspiratory Muscle Training in Critically Ill Patients: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2024 May 26;60(6):869. doi: 10.3390/medicina60060869. PMID 38929486
- [Background] Bissett B, Leditschke IA, Green M, Marzano V, Collins S, Van Haren F. Inspiratory muscle training for intensive care patients: A multidisciplinary practical guide for clinicians. Aust Crit Care. 2019 May;32(3):249-255. doi: 10.1016/j.aucc.2018.06.001. Epub 2018 Jul 11. PMID 30007823
- [Background] Ng DP, Thiviyan P, Shrida S, Ng LWC. Feasibility of Conducting Sit-to-Stand Tests Using Video Consultation. Int J Telemed Appl. 2023 Jul 26;2023:8551680. doi: 10.1155/2023/8551680. eCollection 2023. PMID 39280702
- [Background] Larrateguy S, Otto-Yanez M, Bogado J, Larrateguy L, Barros-Poblete M, Mazzucco G, Blanco I, Gimeno-Santos E, Torres-Castro R. Agreement and Reliability Between Tele-Assessment and In-Person Assessment of the One-Minute Sit-to-Stand Test in Patients with Chronic Respiratory Diseases. J Clin Med. 2025 Jul 16;14(14):5049. doi: 10.3390/jcm14145049. PMID 40725738
- [Background] Salling SL, Jensen JH, Mosegaard SB, Sorensen L, Mechlenburg I. Risk stratification for post-operative pulmonary complications following major cardiothoracic or abdominal surgery: Validation of the PPC Risk Prediction Score for physiotherapist's clinical decision-making. Clin Respir J. 2023 Mar;17(3):229-240. doi: 10.1111/crj.13579. Epub 2023 Jan 3. PMID 36596755
- [Background] Sedlmeier AM, Baumeister SE, Weber A, Fischer B, Thorand B, Ittermann T, Dorr M, Felix SB, Volzke H, Peters A, Leitzmann MF. Relation of body fat mass and fat-free mass to total mortality: results from 7 prospective cohort studies. Am J Clin Nutr. 2021 Mar 11;113(3):639-646. doi: 10.1093/ajcn/nqaa339. PMID 33437985
- [Background] Cao Q, Yu S, Xiong W, Li Y, Li H, Li J, Li F. Waist-hip ratio as a predictor of myocardial infarction risk: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Jul;97(30):e11639. doi: 10.1097/MD.0000000000011639. PMID 30045310
- [Background] Sturgess, T. R., Denehy, L., Tully, E. A., McManus, M., Katijjahbe, M. A., & El-Ansary, D. (2018). The Functional Difficulties Questionnaire: A New Tool for Assessing Physical Function of the Thoracic Region in a Cardiac Surgery Population. Cardiopulmonary Physical Therapy Journal, 29(3), 110-123.
- [Background] Katijjahbe MA, Denehy L, Granger CL, Royse A, Royse C, Logie S, Sturgess T, Md Ali NA, McManus M, Sandy CE, El-Ansary D. Psychometric evaluation of the shortened version of the Functional Difficulties Questionnaire to assess thoracic physical function. Clin Rehabil. 2020 Jan;34(1):132-140. doi: 10.1177/0269215519879476. Epub 2019 Oct 15. PMID 31610700
- [Background] Bowyer AJ, Heiberg J, Sessler DI, Newman S, Royse AG, Royse CF. Validation of the cognitive recovery assessments with the Postoperative Quality of Recovery Scale in patients with low-baseline cognition. Anaesthesia. 2018 Nov;73(11):1382-1391. doi: 10.1111/anae.14402. Epub 2018 Aug 7. PMID 30084176
- [Background] Diab MS, Bilkhu R, Soppa G, Edsell M, Fletcher N, Heiberg J, Royse C, Jahangiri M. The influence of prolonged intensive care stay on quality of life, recovery, and clinical outcomes following cardiac surgery: A prospective cohort study. J Thorac Cardiovasc Surg. 2018 Nov;156(5):1906-1915.e3. doi: 10.1016/j.jtcvs.2018.05.076. Epub 2018 Jun 5. PMID 30336918
- [Background] Zhang X, Tan SS, Fierloos I, Zanutto O, Alhambra-Borras T, Vasiljev V, Bennett S, Rentoumis T, Buranello A, Macchione S, Rouwet E, van Grieken A, Raat H. Evaluation design of the Social Engagement Framework for Addressing the Chronic-disease-challenge (SEFAC): a mindfulness-based intervention to promote the self-management of chronic conditions and a healthy lifestyle. BMC Public Health. 2019 May 30;19(1):664. doi: 10.1186/s12889-019-6979-7. PMID 31146709
- [Background] Bosco E, Hsueh L, McConeghy KW, Gravenstein S, Saade E. Major adverse cardiovascular event definitions used in observational analysis of administrative databases: a systematic review. BMC Med Res Methodol. 2021 Nov 6;21(1):241. doi: 10.1186/s12874-021-01440-5. PMID 34742250
- [Background] Monitoring and Reporting of Safety in Clinical Trials Involving Therapeutic Products and Other Clinical Research Guideline. (2019). Royal Melbourne Hospital: Office for Research.
- [Background] Zhou L, Bao J, Setiawan IMA, Saptono A, Parmanto B. The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11500. doi: 10.2196/11500. PMID 30973342
- [Background] Lalmas, M., O'Brien, H., & Yom-Tov, E. (2015). Measuring User Engagement. Springer International Publishing
- [Background] Junker M, Dunnebeil S, Bohm M, Krcmar H. Usage of a workplace health promotion app: an evaluation of app usage data and medical check-up results. Health Informatics J. 2023 Jan-Mar;29(1):14604582221148058. doi: 10.1177/14604582221148058. PMID 36705467
- [Background] Bauer AM, Iles-Shih M, Ghomi RH, Rue T, Grover T, Kincler N, Miller M, Katon WJ. Acceptability of mHealth augmentation of Collaborative Care: A mixed methods pilot study. Gen Hosp Psychiatry. 2018 Mar-Apr;51:22-29. doi: 10.1016/j.genhosppsych.2017.11.010. Epub 2017 Nov 24. PMID 29272712
- [Background] St-Jules DE, Woolf K, Goldfarb DS, Pompeii ML, Li H, Wang C, Mattoo A, Marcum ZA, Sevick MA. Feasibility and Acceptability of mHealth Interventions for Managing Hyperphosphatemia in Patients Undergoing Hemodialysis. J Ren Nutr. 2021 Jul;31(4):403-410. doi: 10.1053/j.jrn.2020.07.009. Epub 2020 Nov 5. PMID 33160812
- [Background] Hajesmaeel-Gohari S, Khordastan F, Fatehi F, Samzadeh H, Bahaadinbeigy K. The most used questionnaires for evaluating satisfaction, usability, acceptance, and quality outcomes of mobile health. BMC Med Inform Decis Mak. 2022 Jan 27;22(1):22. doi: 10.1186/s12911-022-01764-2. PMID 35081953
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Xue P, Bai AY, Jiang Y, Qiao YL. [WHO global strategy on digital health and its implications to China]. Zhonghua Yu Fang Yi Xue Za Zhi. 2022 Feb 6;56(2):218-221. doi: 10.3760/cma.j.cn112150-20210616-00589. Chinese. PMID 35184452
- [Background] Rivers JT, Smith C, Smith I, Cameron J. The Impact of a Mobile App on Participation in Cardiac Rehabilitation and Understanding Barriers to Success: Comparative Cohort Study. JMIR Cardio. 2022 Jan 17;6(1):e24174. doi: 10.2196/24174. PMID 35037891
- [Background] Waterland JL, Chahal R, Ismail H, Sinton C, Riedel B, Francis JJ, Denehy L. Implementing a telehealth prehabilitation education session for patients preparing for major cancer surgery. BMC Health Serv Res. 2021 May 10;21(1):443. doi: 10.1186/s12913-021-06437-w. PMID 33971869
- [Background] Hughes M, Coolsen MM, Aahlin EK, Harrison EM, McNally SJ, Dejong CH, Lassen K, Wigmore SJ. Attitudes of patients and care providers to enhanced recovery after surgery programs after major abdominal surgery. J Surg Res. 2015 Jan;193(1):102-10. doi: 10.1016/j.jss.2014.06.032. Epub 2014 Jun 23. PMID 25066187
- [Background] Reeve, J., Anderson, L., Raslan, Y., Greeve, C., Ford, J., & Wilson, L. (2019). physiotherapy management of patients undergoing abdominal surgery: A survey of current practice. New Zealand Journal of Physiotherapy, 47(2).
- [Background] Patman S, Bartley A, Ferraz A, Bunting C. Physiotherapy in upper abdominal surgery - what is current practice in Australia? Arch Physiother. 2017 Aug 15;7:11. doi: 10.1186/s40945-017-0039-3. eCollection 2017. PMID 29340205
- [Background] Samnani SS, Umer MF, Mehdi SH, Farid FN. Impact of Preoperative Counselling on Early Postoperative Mobilization and Its Role in Smooth Recovery. Int Sch Res Notices. 2014 Oct 28;2014:250536. doi: 10.1155/2014/250536. eCollection 2014. PMID 27351013
- [Background] Fagevik Olsen M, Wennberg E, Johnsson E, Josefson K, Lonroth H, Lundell L. Randomized clinical study of the prevention of pulmonary complications after thoracoabdominal resection by two different breathing techniques. Br J Surg. 2002 Oct;89(10):1228-34. doi: 10.1046/j.1365-2168.2002.02207.x. PMID 12296888
- [Background] Boden I, Robertson IK, Neil A, Reeve J, Palmer AJ, Skinner EH, Browning L, Anderson L, Hill C, Story D, Denehy L. Preoperative physiotherapy is cost-effective for preventing pulmonary complications after major abdominal surgery: a health economic analysis of a multicentre randomised trial. J Physiother. 2020 Jul;66(3):180-187. doi: 10.1016/j.jphys.2020.06.005. Epub 2020 Jul 14. PMID 32680742
- [Background] Boden I, El-Ansary D, Zalucki N, Robertson IK, Browning L, Skinner EH, Denehy L. Physiotherapy education and training prior to upper abdominal surgery is memorable and has high treatment fidelity: a nested mixed-methods randomised-controlled study. Physiotherapy. 2018 Jun;104(2):194-202. doi: 10.1016/j.physio.2017.08.008. Epub 2017 Sep 1. PMID 28935227
- [Background] Rodriguez-Aldrete D, Candiotti KA, Janakiraman R, Rodriguez-Blanco YF. Trends and New Evidence in the Management of Acute and Chronic Post-Thoracotomy Pain-An Overview of the Literature from 2005 to 2015. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):762-72. doi: 10.1053/j.jvca.2015.07.029. Epub 2015 Jul 29. No abstract available. PMID 26597765
- [Background] Kendall F, Oliveira J, Peleteiro B, Pinho P, Bastos PT. Inspiratory muscle training is effective to reduce postoperative pulmonary complications and length of hospital stay: a systematic review and meta-analysis. Disabil Rehabil. 2018 Apr;40(8):864-882. doi: 10.1080/09638288.2016.1277396. Epub 2017 Jan 17. PMID 28093920
- [Background] Wang YQ, Liu X, Jia Y, Xie J. Impact of breathing exercises in subjects with lung cancer undergoing surgical resection: A systematic review and meta-analysis. J Clin Nurs. 2019 Mar;28(5-6):717-732. doi: 10.1111/jocn.14696. Epub 2018 Nov 20. PMID 30357997
- [Background] Shahood H, Pakai A, Kiss R, Eva B, Szilagyi N, Sandor A, Verzar Z. Effectiveness of Preoperative Chest Physiotherapy in Patients Undergoing Elective Cardiac Surgery, a Systematic Review and Meta-Analysis. Medicina (Kaunas). 2022 Jul 8;58(7):911. doi: 10.3390/medicina58070911. PMID 35888629
- [Background] Xu X, Cheung DST, Smith R, Lai AYK, Lin CC. The effectiveness of pre- and post-operative rehabilitation for lung cancer: A systematic review and meta-analysis on postoperative pulmonary complications and length of hospital stay. Clin Rehabil. 2022 Feb;36(2):172-189. doi: 10.1177/02692155211043267. Epub 2021 Sep 8. PMID 34496658
- [Background] Clode NJ, Perry MA, Wulff L. Does physiotherapy prehabilitation improve pre-surgical outcomes and influence patient expectations prior to knee and hip joint arthroplasty? Int J Orthop Trauma Nurs. 2018 Aug;30:14-19. doi: 10.1016/j.ijotn.2018.05.004. Epub 2018 Jun 25. PMID 29954717
- [Background] Jahic D, Omerovic D, Tanovic AT, Dzankovic F, Campara MT. The Effect of Prehabilitation on Postoperative Outcome in Patients Following Primary Total Knee Arthroplasty. Med Arch. 2018 Dec;72(6):439-443. doi: 10.5455/medarh.2018.72.439-443. PMID 30814777
- [Background] Assouline B, Cools E, Schorer R, Kayser B, Elia N, Licker M. Preoperative Exercise Training to Prevent Postoperative Pulmonary Complications in Adults Undergoing Major Surgery. A Systematic Review and Meta-analysis with Trial Sequential Analysis. Ann Am Thorac Soc. 2021 Apr;18(4):678-688. doi: 10.1513/AnnalsATS.202002-183OC. PMID 33030962
- [Background] Marquina C, Talic S, Vargas-Torres S, Petrova M, Abushanab D, Owen A, Lybrand S, Thomson D, Liew D, Zomer E, Ademi Z. Future burden of cardiovascular disease in Australia: impact on health and economic outcomes between 2020 and 2029. Eur J Prev Cardiol. 2022 May 27;29(8):1212-1219. doi: 10.1093/eurjpc/zwab001. PMID 33686414